CLINICAL TRIAL: NCT02639663
Title: Dental Support Device During Breastfeeding as a Mean for Pain Control
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 559-15-TLV
Record Dates: First submitted 2015-12-21; First posted 2015-12-24 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — Occlusal Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- women whom are interested in breastfeeding and have not begun. (Experimental): Post-partum primi and multiparous women Post-partum primipara and multiparous women whom are interested in breastfeeding and have not begun yet. This arm will be randomized into 2 groups
  1. Intervention group: participants will receive the dental device and be instructed to use it during breastfeeding.
  2. Control group: participants will not receive any device for breastfeeding pain control
  Interventions: Device: dental device
- Post-partum women that have already begun breast feeding (Experimental): 2. Post-partum women that have already begun breast feeding, will receive the dental device and each woman will be serve as her own control (breastfeeding before and after the use of the dental device.
  Interventions: Device: dental device

INTERVENTIONS:
Device: dental device — Leboride
  1. Post-partum primi and multiparous women whom are interested in breastfeeding and have not begun yet. This arm will be randomized into 2 groups
     1. Intervention group: participants will receive the dental device and be instructed to use it during breastfeeding.
     2. Control group: participants will not receive any device for breastfeeding pain control
  2. Post-partum women that have already begun breast feeding, will receive the dental device and each woman will be serve as her own control (breastfeeding before and after the use of the dental device.

SUMMARY:
Leboride is a dental support device that was developed for reducing pain during active labor. It is made of an inert material, placed in the woman's mouth and does not disturb breathing, talking, or any other activity expected during labor. It is a single-use device, each user receives a new one.

This study hypothesis is that the Leboride use can reduce pain during breastfeeding, by that improve women's breastfeeding experience, and increase breastfeeding rates.

DETAILED DESCRIPTION:
Dental support device is effective in increasing isometric force in different muscle contraction [1-7]. In 2009 an avant-garde study [8] found in a small cohort that dental support device during labor, can shorten the second stage and reduce obstetrical interventions such as operative delivery and cesarean section. In this stage the woman has to contract muscles in order to push the fetus through the birth canal.

Leboride is a dental support device that was developed for reducing pain during active labor. It is made of an inert material, placed in the woman's mouth and does not disturb breathing, talking, or any other activity expected during labor. It is a single-use device, each user receives a new one.

This study hypothesis is that the Leboride use can reduce pain during breastfeeding, by that improve women's breastfeeding experience, and increase breastfeeding rates.

ELIGIBILITY:
Inclusion Criteria:

Maternal age 18-45 years. Normal vital signs.

Exclusion Criteria:

Contraindications for breastfeeding. Significant systemic disease that cause pain or require chronic pain relief.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 700 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Rate of change in of the vas scores before and after using this device | 24 months

SECONDARY OUTCOMES:
Duration of breastfeeding | 24 months
The rate of cessation of breastfeeding because of pain | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ariel many, professor, Principal Investigator — Tel Aviv Medical Center

IPD SHARING:
Plan to Share IPD: No